CLINICAL TRIAL: NCT04652479
Title: A Phase 2, Open-Label, Cross-over Study to Assess the Safety and Efficacy of Avexitide in Acquired Hyperinsulinemic Hypoglycemia
Brief Title: Avexitide Safety and Efficacy to Treat Acquired Hyperinsulinemic Hypoglycemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. Tracey McLaughlin, MD (Other)
Collaborators: Eiger BioPharmaceuticals (Industry)
Responsible Party: Principal Investigator, Marilyn Tan, Clinical Assistant Professor of Medicine, Stanford University
Organization: Stanford University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 52880
Record Dates: First submitted 2020-10-27; First posted 2020-12-03 (Actual); Results first posted 2023-06-09 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-05

CONDITIONS: Acquired Hyperinsulinemic Hypoglycemia
Keywords: Post Bariatric Hypoglycemia; avexitide; Post-Bariatric Hypoglycemia; Post-gastrectomy hypoglycemia; Post gastrectomy hypoglycemia; Post-esophagectomy hypoglycemia; Post esophagectomy hypoglycemia; Post-Nissen Fundoplication hypoglycemia; Post Nissen Fundoplication hypoglycemia; Exendin (9-39); Exendin 9-39
MeSH Terms: interventions — exendin (9-39)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Avexitide 45 mg twice daily then avexitide 90 mg once daily (Experimental): Patients will receive one of the two dosing regimens of avexitide for 14 days followed by the other dosing regimen of avextide for 14 days
  Interventions: Drug: Avexitide
- Avexitide 45 mg once daily then avexitide 90 mg twice daily (Experimental): Patients will receive one of the two dosing regimens of avexitide for 14 days followed by the other dosing regimen of avextide for 14 days
  Interventions: Drug: Avexitide

INTERVENTIONS:
Drug: Avexitide — Avexitide (exendin 9-39) is a competitive antagonist of GLP-1 at its receptor

SUMMARY:
The primary goal of this study is to evaluate the safety and efficacy of two different dosing regimens of an investigational drug called Avexitide in treating low blood sugar in patients with Acquired Hyperinsulinemic Hypoglycemia.

ELIGIBILITY:
Inclusion Criteria:

* History of bariatric or upper-gastrointestinal surgery (RYGB, VSG, gastrectomy, esophagectomy, or Nissen fundoplication) at least 12 months prior to the start of Screening
* History of recurrent hypoglycemia occurring after bariatric or upper-GI surgery, as documented in the medical record.
* Body mass index (BMI) of up to 40 kg/m2
* If female, must not be breastfeeding and must have a negative urine pregnancy test result

Exclusion Criteria:

* Major surgery within 6 months before randomization.
* History of or current hyperinsulinism other than Acquired Hyperinsulinism (e.g., insulin autoimmune hypoglycemia).
* Use of agents that may interfere with glucose metabolism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn Tan, MD, Study Director — Stanford University
Locations (1):
- Clinical and Translational Research Unit, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 25 participants entered a 14-day run-in (screening) period during which they wore the continuous glucose monitor (CGM). 17 participants who had at least 2 hypoglycemic events were randomized to a study arm.
Groups:
- Run-in (All Participants): 14-day run-in period during which hypoglycemic events were recorded by CGM.
- Avexitide 45 mg Twice Daily Then Avexitide 90 mg Once Daily; Avexitide 90 mg Once Daily Then Avexitide 45 mg Twice Daily: Patients receive one of the two dosing regimens of avexitide for 14 days followed by the other dosing regimen of avextide for 14 days
Period: Run-in Period (14 Days)
Arm/Group | Run-in (All Participants) | Avexitide 45 mg Twice Daily Then Avexitide 90 mg Once Daily | Avexitide 90 mg Once Daily Then Avexitide 45 mg Twice Daily
Started | 25 | 0 | 0
Completed | 25 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Treatment Period 1 (14 Days)
Arm/Group | Run-in (All Participants) | Avexitide 45 mg Twice Daily Then Avexitide 90 mg Once Daily | Avexitide 90 mg Once Daily Then Avexitide 45 mg Twice Daily
Started | 0 | 8 | 9
Completed | 0 | 8 | 9
Not Completed | 0 | 0 | 0
Period: Washout Period (2 Days)
Arm/Group | Run-in (All Participants) | Avexitide 45 mg Twice Daily Then Avexitide 90 mg Once Daily | Avexitide 90 mg Once Daily Then Avexitide 45 mg Twice Daily
Started | 0 | 8 | 9
Completed | 0 | 8 | 9
Not Completed | 0 | 0 | 0
Period: Treatment Period 2 (14 Days
Arm/Group | Run-in (All Participants) | Avexitide 45 mg Twice Daily Then Avexitide 90 mg Once Daily | Avexitide 90 mg Once Daily Then Avexitide 45 mg Twice Daily
Started | 0 | 8 | 9
Completed Both Interventions With no Major Protocol Deviations | 0 | 8 | 8
Completed | 0 | 8 | 9
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants with no major protocol deviations who were allocated to treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Avexitide 45 mg Twice Daily Then Avexitide 90 mg Once Daily | Avexitide 90 mg Once Daily Then Avexitide 45 mg Twice Daily | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.1 (15.2) | 47.8 (11.2) | 47.9 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 2 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 6 | 7 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 6 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Diurnal Level 2 Hypoglycemia Events (ADA, <54 mg/dL) as Measured by CGM in Patients With Severe Hyperinsulinemic Hypoglycemia (HH)
Description: Level 2 hypoglycemia events (ADA, <54 mg/dL) as measured by CGM and defined as the number of events captured by CGM with glucose measures <54 mg/dL during diurnal hours (8am-10pm) within the run-in period and respective treatment period; for each period data were collected for 14 days, then divided by number of days, then normalized to duration of 14 days.
Time Frame: Run-in period (14 days), treatment period 1 (14 days), and treatment period 2 (14 days)
Population: Participants with no major protocol deviations who were allocated to treatment.
Measure: Mean (Standard Deviation); unit: events per 14 days
Groups:
- Avexitide 45 mg Twice Daily: Patients receive avexitide 45 mg twice daily for 14 days
- Avexitide 90 mg Once Daily: Patients receive avexitide 90 mg once daily for 14 days
Arm/Group | Avexitide 45 mg Twice Daily | Avexitide 90 mg Once Daily
Number analyzed (Participants) | 16 | 16
events per 14 days
  Run-in period | 5.2 (3.52) | 5.2 (3.52)
  Treatment period | 2.7 (2.15) | 2.1 (2.99)
Statistical Analysis 1: Comparison: Avexitide 45 mg Twice Daily; Within-group analysis; Test type: Other; p = 0.0028, Mixed effects model — A p-value of <0.05 would be considered statistically significant
Statistical Analysis 2: Comparison: Avexitide 90 mg Once Daily; Within-group analysis; Test type: Other; p = 0.0005, Mixed effects model — A p-value of <0.05 would be considered statistically significant

2. Secondary Outcome: Rate of Level 2 Hypoglycemia (ADA, <54 mg/dL) as Measured by SMBG
Description: Distinct episodes of Level 2 hypoglycemia (SMBG glucose <54 mg/dL), divided by number of days for run-in period and respective treatment period; for each period data were collected for 14 days, then divided by number of days, then normalized to duration of 14 days.
Time Frame: Run-in period (14 days), treatment period 1 (14 days), and treatment period 2 (14 days)
Population: Participants with no major protocol deviations who were allocated to treatment.
Measure: Mean (Standard Deviation); unit: episodes per 14 days
Arm/Group | Avexitide 45 mg Twice Daily | Avexitide 90 mg Once Daily
Number analyzed (Participants) | 16 | 16
episodes per 14 days
  Run-in period | 2.7 (3.1) | 2.7 (3.1)
  Treatment period | 1.2 (1.4) | 1.3 (3.7)
Statistical Analysis 1: Comparison: Avexitide 45 mg Twice Daily; Within-group analysis; Test type: Other; p = 0.0027, Mixed effects model — A p-value of <0.05 would be considered statistically significant
Statistical Analysis 2: Comparison: Avexitide 90 mg Once Daily; Within-group analysis; Test type: Other; p = 0.0043, Mixed effects model — A p-value of <0.05 would be considered statistically significant

3. Secondary Outcome: Rate of Level 3 Hypoglycemia
Description: Severe events during each treatment period characterized by altered mental and/or physical functioning that requires assistance from another person for recovery; for each period data were collected for 14 days, then divided by number of days, then normalized to duration of 14 days. This would apply regardless of whether a patient actually received external assistance.
Time Frame: Run-in period (14 days), treatment period 1 (14 days), and treatment period 2 (14 days)
Population: Participants with no major protocol deviations who were allocated to treatment.
Measure: Mean (Standard Deviation); unit: events per 14 days
Arm/Group | Avexitide 45 mg Twice Daily | Avexitide 90 mg Once Daily
Number analyzed (Participants) | 16 | 16
events per 14 days
  Run-in period | 2.5 (3.1) | 2.5 (3.1)
  Treatment period | 0.8 (1.2) | 0.9 (2.9)
Statistical Analysis 1: Comparison: Avexitide 45 mg Twice Daily; Within-group analysis; Test type: Other; p = 0.0003, Mixed effects model — A p-value of <0.05 would be considered statistically significant
Statistical Analysis 2: Comparison: Avexitide 90 mg Once Daily; Within-group analysis; Test type: Other; p = 0.0003, Mixed effects model — A p-value of <0.05 would be considered statistically significant

4. Secondary Outcome: Percent Time in Level 2 Hypoglycemia (<54 mg/dL) as Measured by CGM (Diurnal Time)
Description: Percentage of time in level 2 hypoglycemia (<54mg/dL by CGM) during diurnal hours (8am-10pm) within the run-in period and respective treatment period; for each period data were collected for 14 days, then divided by number of days, then normalized to duration of 14 days.
Time Frame: Run-in period (14 days), treatment period 1 (14 days), and treatment period 2 (14 days)
Population: Participants with no major protocol deviations who were allocated to treatment.
Measure: Mean (Standard Deviation); unit: percentage of time per 14 days
Arm/Group | Avexitide 45 mg Twice Daily | Avexitide 90 mg Once Daily
Number analyzed (Participants) | 16 | 16
percentage of time per 14 days
  Run-in period | 1.50 (1.32) | 1.50 (1.32)
  Treatment period | 0.96 (0.74) | 0.48 (0.82)
Statistical Analysis 1: Comparison: Avexitide 45 mg Twice Daily vs Avexitide 90 mg Once Daily; Between-group analysis of change from baseline; Test type: Other; p = 0.161, t-test, 2 sided — A p-value of <0.05 would be considered statistically significant
Statistical Analysis 2: Comparison: Avexitide 45 mg Twice Daily; Within-group analysis of change from baseline; Test type: Other; p = 0.201, t-test, 2 sided — A p-value of <0.05 would be considered statistically significant; Mean Difference (Net) = -35.66
Statistical Analysis 3: Comparison: Avexitide 90 mg Once Daily; Within-group analysis of change from baseline; Test type: Other; p = 0.001, t-test, 2 sided — A p-value of <0.05 would be considered statistically significant; Mean Difference (Net) = -67.65

5. Secondary Outcome: Percent Time in Level 1 Hypoglycemia (<70 mg/dL) as Measured by CGM (Diurnal Time)
Description: Percentage of time in level 1 hypoglycemia (<70mg/dL by CGM) during diurnal hours (8am-10pm) within the run-in period and respective treatment period; for each period data were collected for 14 days, then divided by number of days, then normalized to duration of 14 days.
Time Frame: Run-in period (14 days), treatment period 1 (14 days), and treatment period 2 (14 days)
Population: Participants with no major protocol deviations who were allocated to treatment.
Measure: Mean (Standard Deviation); unit: percentage of time per 14 days
Arm/Group | Avexitide 45 mg Twice Daily | Avexitide 90 mg Once Daily
Number analyzed (Participants) | 16 | 16
percentage of time per 14 days
  Run-in period | 4.20 (2.75) | 4.20 (2.75)
  Treatment period | 2.86 (1.54) | 1.96 (1.63)
Statistical Analysis 1: Comparison: Avexitide 45 mg Twice Daily vs Avexitide 90 mg Once Daily; Between-group analysis of change from baseline; Test type: Other; p = 0.145, t-test, 2 sided — A p-value of <0.05 would be considered statistically significant
Statistical Analysis 2: Comparison: Avexitide 45 mg Twice Daily; Within-group analysis of change from baseline; Test type: Other; p = 0.111, t-test, 2 sided — A p-value of <0.05 would be considered statistically significant; Mean Difference (Net) = -31.88 — Change in percentage
Statistical Analysis 3: Comparison: Avexitide 90 mg Once Daily; Within-group analysis of change from baseline; Test type: Other; p = 0.001, t-test, 2 sided — A p-value of <0.05 would be considered statistically significant; Mean Difference (Net) = -53.37 — Change in percentage

6. Secondary Outcome: Postprandial Glycemia During Standardized Mixed Meal Consumption
Description: Change from Baseline in glycemia During Standardized Mixed Meal Consumption
Time Frame: 3 Hours Following Standardized Liquid Meal
Population: Data were not collected for this outcome
Arm/Group | Avexitide 45 mg Twice Daily | Avexitide 90 mg Once Daily
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 44 days
Groups:
- Run-in Period: Adverse events collected during the run-in period
- Avexitide 45 mg Twice Daily: Adverse events collected during the avexitide 45 mg twice daily treatment period
- Avexitide 90 mg Once Daily: Adverse events collected during the avexitide 90 mg once daily treatment period
Arm/Group | Run-in Period | Avexitide 45 mg Twice Daily | Avexitide 90 mg Once Daily
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/25 | 7/17 | 8/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Run-in Period (N=25) | Avexitide 45 mg Twice Daily (N=17) | Avexitide 90 mg Once Daily (N=17)
injection site bruising (Skin and subcutaneous tissue disorders) | 0 (0) | 6 (6) | 8 (8)
loose stools (Gastrointestinal disorders) | 0 (0) | 5 (5) | 4 (4)
headache (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-13): https://cdn.clinicaltrials.gov/large-docs/79/NCT04652479/Prot_SAP_000.pdf